CLINICAL TRIAL: NCT04025437
Title: Neoadjuvant Radiotherapy for Patients With Hepatocellular Carcinoma Involving Type I Portal Vein Tumor Thrombus
Brief Title: Neoadjuvant Radiotherapy for HCC Involving Type I PVTT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT-HCC-PVTT
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Neoadjuvant Radiotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatectomy alone (Experimental): Patients in this group will receive hepatectomy alone.
  Interventions: Procedure: Hepatectomy alone
- Neoadjuvant radiotherapy plus hepatectomy (Active Comparator): Radiotherapy for type I PVTT will be perfomed before hepatectomy. Hepatic resection will be performed in about 4 weeks after radiotherapy.
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Procedure: Hepatectomy alone — Patients in this group will receive hepatectomy alone.
  Arms: Hepatectomy alone
Radiation: Neoadjuvant radiotherapy — Radiotherapy for type I PVTT will be perfomed before hepatectomy. Hepatic resection will be performed in about 4 weeks after radiotherapy.
  Arms: Neoadjuvant radiotherapy plus hepatectomy

SUMMARY:
The rate of patients with hepatocellular carcinoma (HCC) involving portal vein tumor thrombus (PVTT) is up to 50% in Guangxi province, China. Some of them will receive hepatic resection, especially those with type I or II PVTT. However, 5-years recurrence rate is up to 75% after surgery. Some retrospective studies found postoperative radiotherapy may reduce the rate of recurrence. Moreover, few retrospective studies also found neoadjuvant radiotherapy (PMID: 27317960) may improve overall survival for HCC patients involving type II/III PVTT. However, the safety and efficacy of neoadjuvant raidotherapy for HCC involving type I PVTT is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;
* Patients with resectable primary hepatocellular carcinoma and Cheng's type I portal vein tumor thrombus;
* Child-Pugh A or B (7 score) liver function;
* With more than 3 months expected survival;
* The volume of residual liver more than 30%;
* Patients agree to take part in.

Exclusion Criteria:

* Patients with primary hepatocellular carcinoma and Cheng's type II/III/IV portal vein tumor thrombus
* Previous history of epigastric radiotherapy
* With extrahepatic metastasis
* With radiotherapy contraindication;
* Pregnant woman or sucking period;
* With repture tumor;
* With other cancer in previous five years;
* With chemothrapy, target therapy or immunosuppressive drugs therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  From the date of hepatectomy or neoadjuvant radiotherapy to death or the end of follow-up.

SECONDARY OUTCOMES:
Recurrence-free survival | 1 year
  From the date of hepatectomy to HCC recurrence or the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Zhong Tang, MD, Study Director — Cancer Hospital of Guangxi Medical University
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon SM, Ryoo BY, Lee SJ, Kim JH, Shin JH, An JH, Lee HC, Lim YS. Efficacy and Safety of Transarterial Chemoembolization Plus External Beam Radiotherapy vs Sorafenib in Hepatocellular Carcinoma With Macroscopic Vascular Invasion: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):661-669. doi: 10.1001/jamaoncol.2017.5847. PMID 29543938
- [Background] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690
- [Background] Kudo M, Ueshima K, Yokosuka O, Ogasawara S, Obi S, Izumi N, Aikata H, Nagano H, Hatano E, Sasaki Y, Hino K, Kumada T, Yamamoto K, Imai Y, Iwadou S, Ogawa C, Okusaka T, Kanai F, Akazawa K, Yoshimura KI, Johnson P, Arai Y; SILIUS study group. Sorafenib plus low-dose cisplatin and fluorouracil hepatic arterial infusion chemotherapy versus sorafenib alone in patients with advanced hepatocellular carcinoma (SILIUS): a randomised, open label, phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):424-432. doi: 10.1016/S2468-1253(18)30078-5. Epub 2018 Apr 7. PMID 29631810
- [Background] Li N, Feng S, Xue J, Wei XB, Shi J, Guo WX, Lau WY, Wu MC, Cheng SQ, Meng Y. Hepatocellular carcinoma with main portal vein tumor thrombus: a comparative study comparing hepatectomy with or without neoadjuvant radiotherapy. HPB (Oxford). 2016 Jun;18(6):549-56. doi: 10.1016/j.hpb.2016.04.003. Epub 2016 May 7. PMID 27317960